CLINICAL TRIAL: NCT04990453
Title: PEEK Versus Metallic Framework for Extra Coronal Attachment Mandibular Bilateral Distally Extension Removable Partial Denture- Evaluation of Abutments Bone Height Changes and Patient Satisfaction. A Randomized Clinical Trial.
Brief Title: PEEK Versus Metallic Framework for Extra Coronal Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nourhan Ahmed Ragheb, Lecturer , Prosthodontist, Department of Prosthodontics, Faculty of Oral & Dental Medicine,Kafr El-shiekh University, Kafr El-shiekh ,Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KD/12/21
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Removable Partial Denture
Keywords: Framework materials; Removable partial denture; Patient satisfaction; PEEK; Bone changes
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPD frameworks fabricated from PEEK material (Other): 14 patients received extracoronal precision attachment RPD frameworks fabricated from PEEK material using milling machine (CAD/CAM technology)
  Interventions: Other: RPD frameworks fabricated from PEEK material
- RPD frameworks fabricated from Co-Cr (Other): 14 patients received extracoronal precision attachment RPD frameworks fabricated from Co-Cr material using casting machine
  Interventions: Other: RPD frameworks fabricated from PEEK material

INTERVENTIONS:
Other: RPD frameworks fabricated from PEEK material — extracoronal precision attachment RPD frameworks fabricated from PEEK material using milling machine (CAD/CAM technology)

SUMMARY:
Purpose: The present study was aimed to evaluate the bone height changes around abutments with two different framework materials for extracoronal attachment mandibular bilateral distally extension removable partial denture (RPD) and compare patient satisfaction associated with its use.

Materials and methods:

Ten partially edentulous patients (long span kennedy class I) were selected, for all patients splinting of remaining abutment were done by porcelain fused to metal bridges, after cementation the RPD frameworks were digitally designed by CAD software and printed into 3-D resin pattern after intra-oral try in of these patterns, the patients were divided into two equalized groups, the patients in first group received extracoronal attachment (RPD)with from milled PEEK (Juvora) framework. While patients in second group received extracoronal attachment (RPD) with conventional metal framework by lost wax technique. Digital radiography was used for bone height assessment of distal abutment at time of prosthesis insertion, 6 and 12 months later. Patient satisfaction was measured using VAS scale.

DETAILED DESCRIPTION:
I-Patient selection For this study, ten patients (50-60) with mean age 55 years will be selected from out clinic patients Prosthodontic Department, Faculty of Dentistry, Kafr El_Sheikh University. The patients will have the following inclusion criteria:- Completely edentulous maxillary arch against partially edentulous mandible with only remaining mandibular anterior teeth. The selected patients will be free from any systemic diseases, the patients have Angle class I maxillomandibular skeletal relation, the distal extension ridge will be well formed and covered by healthy, firm mucosa, Good abutments with healthy periodontal ligament and suitable crown/root ratio (CRR) as verified by periapical radiograph.

The exclusion criteria to the patients were:

Patients with any systemic disease that could affect the rate of bone resorption which verified by obtaining a medical history, Patients with Para-functional habits (Bruxism and clenching), Patients with any septic foci or impacted teeth as verified by panoramic radiograph, Patients with tilted or rotated abutments. Patients with soft tissue undercuts involved in the design.

For every patient the following procedures were done:

1. Diagnostic Digital panoramic X-ray will be done, then Diagnostic Long Cone standard Digital peri-apical radiographs for canines will be taken to determine crown /root ratio.
2. Scaling and/or root planning for remaining mandibular anterior teeth will be carried out, follow up of good oral hygiene measures before start of treatment plan for one month
3. Correction of irregular occlusal plane will be done either by enameloplasty for overerupted teeth or restoration by adding composite for infraerupted one if needed.
4. All selected patients in this study will be informed about all procedures that will be done and the need for regular and frequent recalls. All patients will sign the consent form of ethical committee in Faculty of dentistry, Kafr El_Sheikh university.

II. Prosthetic procedures:

For each patient, the definitive mandibular extra coronal attachment removable partial denture will be designed using CAD/CAM technology

-Scanning the Master Model The mandibular master cast with porcelain crowns will be then fixed on the scanner table and scanned using the 3D scanner to obtain the standard triangulation file (STL) format.

(Master cast) will be fixed on the table of 3 Shape scanning machine dental system, after application of scan-able spray (Telescan Spray zur vorbereitong von oberflacohen .Teleskop kronen) over the stone teeth and porcelain crowns of master model.

* Digital process and CAD Design of Removable Partial Denture Frameworks Secondary surveying of the virtual master cast will be performed digitally according to the predetermined path of insertion which will be used
* STL file of the virtual framework will be used to print the resin pattern using 3D printer which checked on the master cast before intraoral try in. (A tentative resin frameworks will be constructed by utilizing rapid prototyping technique to examine the accuracy of the framework)
* Intraoral try in will be done to verify all the framework components and determine any needed corrections that would be done on the STL file.
* Framework construction:

According to the framework material and technique of construction, the patients will be equally divided in to two groups as the following:

Group A: Patients will receive RPD frameworks fabricated from PEEK material using milling machine (CAD/CAM technology).

Group B: Patients will receive RPD frameworks fabricated from Co-Cr material using casting machine.

For group (A) PEEK RPD framework construction will be done as follow:

The virtual 3D framework (STL) file will be sent to the milling machine to begin the milling process of PEEK discs to produce mandibular attachment removable partial denture PEEK framework.

The PEEK framework will be then finished and polished then reseated on the master cast to check its fitting. After that, the PEEK framework will be tried in the patient mouth to check its fitting.

For group (B) metallic RPD framework construction was done as follow:

The virtual 3D framework (STL) file with supporting bars and sprues will be printed with resin and then invested, burnt out, and casted with chromium cobalt alloy to produce mandibular attachment removable partial denture metallic framework.

The metallic RPD framework will be then finished, polished and reseated on the master cast to check its adaptation. After that, the metallic framework will be tried in the patient mouth to check its fitting.

For each patient the in the two groups:

1. Maxillary auto polymerized resin special tray will be constructed.
2. Altered cast impression technique will be made Record blocks were constructed on maxillary secondary cast and mandibular framework on the altered master cast.
3. After registration of the jaw relation, the casts will be mounted on semi-adjustable articulator using maxillary face bow for mounting maxillary cast and centric inter-occlusal record for mandibular one.
4. Semi-anatomic maxillary posterior teeth will be arranged against flat mandibular teeth to achieve balanced lingualized occlusion.
5. After try-in in the patient mouth, the denture will be processed and the occlusion was refined.
6. Matrix inserting instrument will be used to insert and push the matrix with desired friction in its place (green plastic matrix for light snap in friction was the selected matrix), and functional pick up will be done during cementaion of crowns by applying finger pressure during setting of cement with proper orientation provided by the two temporary indirect retainers.
7. All crowns will be cemented by resin luting cement during insertion of the extracoronal precision attachment removable partial denture.
8. Periapical radiographs of abutment teeth and implant will be taken and digital panoramic radiographs will be made at the time of insertion and after 6 and 12 months later

ELIGIBILITY:
Inclusion Criteria:

* The average age of selected patients was from 55 -60 years .

  * Completely edentulous maxillary arch opposed by partially edentulous mandible with only remaining mandibular anterior teeth.
  * All selected patients were free from any systemic diseases,
  * All patients had Angle class I maxillomandibular skeletal relation,
  * The distal extension ridge was well formed and covered by healthful, firm mucosa,
  * Suitable abutments with healthy periodontal ligament and appropriate crown/root ratio (CRR) as verified by periapical radiograph.

The exclusion criteria to the patients were:

* patients with any systemic disease that could affect the rate of bone resorption which confirmed by obtaining a medical history,
* Patients with Para-functional habits (Bruxism and clenching),
* Patients with any septic foci or impacted teeth as proved by panoramic radiograph,
* Patients with tilted or rotated abutments. Patients with soft tissue undercuts had involved in the design.

Ages: 55 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
evaluation of bone height changes | 12 months
  An image plate was attached on a radiographic stent specially constructed for each patient to made a standardized periapical radiograph for the abutments by using the Dentsply/rinn XCP tools (long, round BID cone paralleling technique) according to:
  Image analysis:
  The linear measurement system contributed by the special software of the Vista-scan machine was used for measuring the mesial and distal marginal bone height around the canine abutments bilaterally in both groups.

SECONDARY OUTCOMES:
Patient satisfaction (VAS) | 12 months
  Patient satisfaction was assessed using a questionnaire based on visual analog scale (VAS). Satisfaction after six months follow up period was tested concerning comfort, esthetics, stability, speaking retention, general satisfaction. Patients were requested to mark their answer (amount of satisfaction) on a 100-mm line (with zero indicates to not satisfied at all and 100 indicates to completely satisfied). Higher VAS scores showed high satisfaction and lower scores indicated low satisfaction. The mean of the answers (length of the lines from zero to the marks in mm) for every question was subjected to statistical analysis.
  All dimensions of this instrument are highly associated with the items of general satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral & Dental Medicine,Kafr El-shiekh University, Kafr El-shiekh ,Egypt, Kafr El-shiekh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol